CLINICAL TRIAL: NCT01137877
Title: Growth and Tolerance of Healthy Term Infants to a New Infant Formula
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The control product was recalled.
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie Swearengin, Director Clinical Research Operations, Abbott Nutrition
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK66
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Healthy Term Infants
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Infant Formula #1 (Active Comparator): Milk-based Infant Formula Powder
  Interventions: Other: Milk based infant formula powder
- Investigational Infant Formula #1 (Experimental): Investigational Milk-based Infant Formula Powder
  Interventions: Other: Investigational Infant Formula #1
- Investigational Infant Formula #2 (Experimental): Investigational Milk based infant formula powder
  Interventions: Other: Investigational Infant Formula #2
- Human Milk (Active Comparator): Reference group
  Interventions: Other: Human Milk

INTERVENTIONS:
Other: Milk based infant formula powder — milk based infant formula ad lib
  Arms: Infant Formula #1
Other: Investigational Infant Formula #1 — Milk based infant formula ad lib
  Arms: Investigational Infant Formula #1
Other: Investigational Infant Formula #2 — Milk based infant formula powder ad lib
  Arms: Investigational Infant Formula #2
Other: Human Milk — Human milk ad lib
  Arms: Human Milk

SUMMARY:
The objective of this study is to evaluate the effect of two experimental milk-based infant formulas on the growth and gastrointestinal (GI) tolerance of term infants.

ELIGIBILITY:
Inclusion Criteria:

* in good health
* singleton full term birth
* Birth weight > 2490 g.
* Infant is between 0 and 11 days of age
* Infants using medications , home remedies , herbal preparations, prebiotics, probiotics or rehydration fluids that might affect GI tolerance
* If formula-fed, parent(s) confirm their intention to feed their infant the study product as the sole source of nutrition for the duration of the study
* If human milk-fed, parent(s) confirm their intention to feed their infant human milk as the sole source of nutrition
* not consuming vitamin or mineral supplements, solid foods or juices through the duration of the study

Exclusion Criteria:

adverse maternal, fetal or infant medical history with potential for effects on tolerance, growth, and/or development.

Ages: 1 Day to 11 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 399 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
weight gain | 14 to 119 days of age

SECONDARY OUTCOMES:
GI tolerance | 14 to 119 days of age
anthropometrics | 14 to 119 days of age

CONTACTS AND LOCATIONS:
Overall Officials: Timberly Williams, PhD, Study Chair — Abbott Nutrition
Locations (20):
- United States (20):
  - Arkansas Children's Hospital Research, Little Rock, Arkansas
  - Facey Medical Foundation, Mission Hills, California
  - Norwich Pediatric Group, Norwich, Connecticut
  - All Women's Healthcare of West Broward, Inc, Plantation, Florida
  - SCORE Physician Alliance LLC, St. Petersburg, Florida
  - USF College of Medicine, USF Health, Department of Pediatrics, Tampa, Florida
  - Northpoint Pediatrics, Indianapolis, Indiana
  - University of Louisville Department of Pediatrics, Louisville, Kentucky
  - New England Center for Clinical Research, Inc, Fall River, Massachusetts
  - Wayzata Children's Clinic Ridgeview Research, Chaska, Minnesota
  - Midwest Children's Health Research Institute, LLC, Lincoln, Nebraska
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Cary Pediatric Center, Cary, North Carolina
  - Dayton Clinical Research, Dayton, Ohio
  - Ohio Pediatric Research Association, Inc, Huber Heights, Ohio
  - Parma Pediatrics, Parma, Ohio
  - Comprehensive Pediatrics, Inc, Westlake, Ohio
  - Sanford Clinic Family Medicine 34th and Kiwanis, Sioux Falls, South Dakota
  - DCOL Center for Clinical Research, Longview, Texas
  - Rockwood Clinic North Pediatrics, Spokane, Washington